CLINICAL TRIAL: NCT02985905
Title: The Effect of Oral Zinc Supplementation on Thiol Oxido-reductive Index and Thiol Related Enzymes in Spermatozoa of Iraqi Asthenospermic Patients
Brief Title: The Effect of Oral Zinc Supplementation on Thiol Oxido-reductive Index
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: mahmoud hussein hadwan (Other)
Collaborators: Ministry of Health, Iraq (Network)
Responsible Party: Sponsor-Investigator, mahmoud hussein hadwan, Principal Investigator, Babylon University
Organization: Babylon University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Babil-4
Record Dates: First submitted 2016-12-02; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Asthenozoospermia
Keywords: Zinc supplementation; Thiol; Glutathione peroxidase; Sulfhydryl oxidase
MeSH Terms: conditions — Asthenozoospermia | interventions — Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zinc sulfate (Experimental): 60 subfertile (age 32.5±3.23 year) men with asthenozoospermia was treated with zinc sulfate,every participant took two capsules of zinc sulfate per day for three months (each one 220 mg).
  Interventions: Dietary Supplement: zinc sulfate
- Healthy control (No Intervention): 60 fertile (age 31.6±3.3 year) men, no treatment

INTERVENTIONS:
Dietary Supplement: zinc sulfate — The subfertile group treated with zinc sulfate, every participant took two capsules of zinc sulfate per day for three months (each one 220 mg).
  Arms: Zinc sulfate

SUMMARY:
Although several studies have considered the relationship between infertility and semen thiol compounds levels, no study on the effects of asthenospermia treatments such as oral zinc supplementation on thiol related enzymes activity which are important in fertility of the individual has been reported.

DETAILED DESCRIPTION:
The present study was conducted to study the effect of zinc supplementation on the quantitative and qualitative characteristics of semen along with reduced thiol, oxidized thiol and thiol related enzymes in the seminal plasma of asthenospermic patients.

ELIGIBILITY:
Inclusion Criteria:

* The presence of asthenozoospermia in the semen sample.

Exclusion Criteria:

* The absence of endocrinopathy, varicocele, and female factor infertility. Smokers and alcoholic men were excluded from the study because of their recognized high seminal ROS levels and decreased antioxidant levels.

Ages: 26 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Thiol oxido-reductive index levels in spermatozoa and seminal plasma. The investigators evaluated the effects of zinc sulfate (220 mg/d) supplementation on Thiol oxido-reductive index levels. | up to three months.

SECONDARY OUTCOMES:
Glutathione peroxidase activity levels in spermatozoa and seminal plasma. The investigators evaluated the effects of zinc sulfate (220 mg/d) supplementation on Glutathione peroxidase activity levels. | up to three months.
Sulfhydryl oxidase activity levels in spermatozoa and seminal plasma. The investigators evaluated the effects of zinc sulfate (220 mg/d) supplementation on Sulfhydryl oxidase activity levels. | up to three months.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Hadwan, PhD, Principal Investigator — Babylon University; L Almashhedy, PhD, Study Director — Babylon University; Alsalman Abdulrrazaq, PhD, Study Chair — Babylon University
Locations (1):
- Mahmoud Hadwan, Hillah, Babylon, Iraq

IPD SHARING:
Plan to Share IPD: Yes
I plan to publish the results in a scientific journal

REFERENCES:
- [Derived] Alsalman ARS, Almashhedy LA, Hadwan MH. Effect of Oral Zinc Supplementation on the Thiol Oxido-Reductive Index and Thiol-Related Enzymes in Seminal Plasma and Spermatozoa of Iraqi Asthenospermic Patients. Biol Trace Elem Res. 2018 Aug;184(2):340-349. doi: 10.1007/s12011-017-1215-8. Epub 2017 Dec 8. PMID 29222649